CLINICAL TRIAL: NCT04003051
Title: Mobile Delivery of a Coping and Adherence Program for Head and Neck Cancer Patients Being Treated in Community Care Settings
Brief Title: Web-Based Program in Helping Patients With Head and Neck Cancer Adhere to Swallowing Exercises and Coping Strategies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-1022; NCI-2019-01687 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1022 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Throat Carcinoma
Keywords: Head and neck cancer; swallowing; trismus; adherence; coping; rural; website; access
MeSH Terms: conditions — Head and Neck Neoplasms; Trismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Project Prepare website) (Experimental): Patients use the password-protected Project Prepare website on a computer, tablet, or phone over 10 weeks to view: videos of the swallowing and trismus exercises, tips and stories from former patients, what to expect each week of treatment, recipes and cooking demonstrations, how to take care of their teeth during treatment, strategies for stress relief, and strategies for dry mouth and nausea. This website is designed to reach underserved populations who do not have ready access to specialized preventive care.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Use Project Prepare website
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well a web-based program called Project Prepare works in helping patients with head and neck cancer adhere to swallowing and trismus exercises and coping strategies. Head and neck cancer patients who receive radiation therapy are at risk for permanent swallowing disorders and other side effects. Because of these potential problems, swallowing exercises and coping strategies are important parts of recovery. A web-based program designed to increase adherence to preventive exercises may help patients with head and neck cancer ameliorate the long-term effects of radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the impact of a web-based adherence program (PREPARE) on self-reported swallowing function in head and neck cancer patients during radiation.

SECONDARY OBJECTIVE:

I. To determine community participant adherence to targeted swallowing and trismus exercises delivered by the PREPARE website video demonstrations.

EXPLORATORY OBJECTIVE:

I. To promote the long-term dissemination of the Dysphagia Prevention program through measurement of patient satisfaction and engagement metrics, training and continual feedback between the MD Anderson Cancer Center (MDACC) research site and community collaborative research sites.

OUTLINE:

Patients use the password-protected Project Prepare website on a computer, tablet, or phone over 10 weeks to view: videos of the swallowing and trismus exercises, tips and stories from former patients, what to expect each week of treatment, recipes and cooking demonstrations, how to take care of their teeth during treatment, strategies for stress relief, and strategies for dry mouth and nausea. This website is designed to reach underserved populations who do not have ready access to specialized preventive care.

After completion of study, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Receiving radiation treatment with curative intent for throat cancer
* Can read and speak English or Spanish well enough to answer our questionnaires and understand our website content.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in self-reported swallowing function | Baseline up to 6 months post-radiation
  Assessed with the MD Anderson Dysphagia Inventory (MDADI). Will first test for changes in self-reported swallowing function outcome with the MDADI between baseline and follow-up using one-tailed paired t-tests. Correlations and multivariate analyses regressing self-reported adherence to exercises against self-reported swallowing function will be analyzed similarly and appropriately.

SECONDARY OUTCOMES:
Website usage data | Up to 6 months post-radiation
  Piwik analytics will be used to record usage data regarding patient engagement with the website (e.g. whether the patient looked at the website that week, number of minutes and number of navigations and pages visited).

CONTACTS AND LOCATIONS:
Overall Officials: Eileen H Shinn, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Texas Health Care-Otolaryngology and Plastic Surgery Associates, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org